CLINICAL TRIAL: NCT02079246
Title: An Open-label Extension Study to Evaluate the Long-term Safety and Tolerability of Idalopirdine (Lu AE58054) as Adjunctive Treatment to Donepezil in Patients With Mild-moderate Alzheimer's Disease
Brief Title: Long-term Safety and Tolerability of Idalopirdine (Lu AE58054) as Adjunctive Treatment to Donepezil in Patients With Mild-moderate Alzheimer's Disease
Acronym: STAR Extension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14861B; 2013-000001-23 (EudraCT Number)
Record Dates: First submitted 2014-02-28; First posted 2014-03-05 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — (2-(6-fluoro-1H-indol-3-yl)-ethyl)-(3-(2,2,3,3-tetrafluoropropoxy)benzyl)amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Idalopirdine (Lu AE58054) 60 mg (Experimental): Idalopirdine 60 mg adjunct to 10 mg donepezil. The dose of idalopirdine could be decreased from 60 mg to 30 mg if 60 mg was not well tolerated. The dose of donepezil was to be maintained throughout the study.
  Interventions: Drug: Idalopirdine 60 mg
- Idalopirdine 60 mg + memantine (Experimental): Idalopirdine 60 mg as adjunct to 10 mg donepezil and memantine (patient's individualised maintenance dose, either immediate-release (IR) 20 mg/day (recommended target dose) or extended release (XR) 28 mg/day (recommended target dose). Memantine was administered to approximately 100 patients included in the OLEX-MEM. The dose of idalopirdine could be decreased from 60 mg to 30 mg if 60 mg was not well tolerated. The dose of donepezil was to be maintained throughout the study. The dose of memantine could be changed at any time throughout the study.
  Interventions: Drug: Idalopirdine 60 mg

INTERVENTIONS:
Drug: Idalopirdine 60 mg — once daily, encapsulated tablets, orally

SUMMARY:
To evaluate the long-term safety and tolerability of idalopirdine (Lu AE58054) as adjunctive therapy to donepezil in patients with mild-moderate Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
This is an interventional, multi-national, multi-site, open-label extension study in patients with mild to moderate AD who completed the 24-week lead-in study 14861A (NCT01955161) or 14862A (NCT02006641).

Patients received 28-weeks of open-label treatment with idalopirdine 60 mg/day (option to reduce to 30 mg/day) as adjunctive treatment to donepezil. Approximately 100 patients, who had completed the initial 28-week period (OLEX), were included in a 24 week open-label treatment period with memantine (OLEX-MEM) that evaluated the safety and tolerability of concomitant memantine therapy in patients who were already on a stable treatment with idalopirdine and donepezil and for whom memantine treatment was clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* the patient has completed Visit 7 (Completion Visit) in the lead-in double-blind, placebo controlled clinical studies 14861A/NCT01955161 or 14862A/NCT02006641

For patients in the OLEX-MEM:

* The patient has completed Visit 6 (Week 28) of the OLEX.
* The patient, according to the judgement of the investigator, requires initiation of treatment with memantine as per local label/SmPC/treatment guidelines.

Exclusion Criteria:

* The patient has a moderate or severe ongoing adverse event from the lead-in study considered a potential safety risk by the investigator.
* The patient has experienced seizures before Completion Visit in the lead-in study.
* The patient has evidence of clinically significant disease.
* The patient's donepezil treatment is likely to be interrupted or discontinued during the study.
* The patient is receiving therapy with another acetylcholinesterase inhibitors (AChEI).

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1463 (Actual)
Dates: Start 2014-04-07 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (258):
- United States (64):
  - US027, Birmingham, Alabama
  - US012, Phoenix, Arizona
  - US338, Phoenix, Arizona
  - US024, Little Rock, Arkansas
  - US351, Carlsbad, California
  - US346, Costa Mesa, California
  - US327, Fullerton, California
  - US023, Imperial, California
  - US045, Long Beach, California
  - US307, Redlands, California
  - US058, San Francisco, California
  - US018, Santa Ana, California
  - US301, Santa Rosa, California
  - US021, Bradenton, Florida
  - US050, Brooksville, Florida
  - US308, Delray Beach, Florida
  - US320, Hallandale, Florida
  - US347, Hialeah, Florida
  - US340, Lake Worth, Florida
  - US303, Miami, Florida
  - US313, Miami, Florida
  - US345, Orange City, Florida
  - US019, Orlando, Florida
  - US309, Palm Beach Gardens, Florida
  - US038, Port Charlotte, Florida
  - US302, Sunrise, Florida
  - US304, Atlanta, Georgia
  - US360, Augusta, Georgia
  - US048, Kailua, Hawaii
  - US030, Chicago, Illinois
  - US040, Indianapolis, Indiana
  - US334, Lake Charles, Louisiana
  - US036, Freeport, Maine
  - US344, Boston, Massachusetts
  - US035, Kalamazoo, Michigan
  - US310, Saint Paul, Minnesota
  - US041, Flowood, Mississippi
  - US321, Hattiesburg, Mississippi
  - US339, Paterson, New Jersey
  - US046, Princeton, New Jersey
  - US028, Toms River, New Jersey
  - US044, Toms River, New Jersey
  - US014, Manhasset, New York
  - US029, New York, New York
  - US312, Staten Island, New York
  - US316, Charlotte, North Carolina
  - US336, Winston-Salem, North Carolina
  - US007, Centerville, Ohio
  - US323, Cincinnati, Ohio
  - US006, Columbus, Ohio
  - US306, Columbus, Ohio
  - US352, Lakewood, Ohio
  - US333, Oklahoma City, Oklahoma
  - US026, Portland, Oregon
  - US057, Jenkintown, Pennsylvania
  - US324, Pittsburgh, Pennsylvania
  - US341, Pittsburgh, Pennsylvania
  - US319, Port Royal, South Carolina
  - US356, Cordova, Tennessee
  - US343, Fort Worth, Texas
  - US354, Houston, Texas
  - US047, Arlington, Virginia
  - US025, Madison, Wisconsin
  - US004, Milwaukee, Wisconsin
- Argentina (20):
  - AR303, Banfield
  - AR007, Buenos Aires
  - AR312, Buenos Aires
  - AR003, Ciudad Autonoma Buenos Aires
  - AR304, Ciudad Autonoma Buenos Aires
  - AR308, Ciudad Autonoma Buenos Aires
  - AR311, Ciudad Autonoma Buenos Aires
  - AR313, Ciudad Autonoma Buenos Aires
  - AR314, Ciudad Autonoma Buenos Aires
  - AR009, Córdoba
  - AR307, Córdoba
  - AR309, Córdoba
  - AR305, Godoy Cruz
  - AR004, Mar del Plata
  - AR005, Mendoza
  - AR008, Mendoza
  - AR310, Mendoza
  - AR010, Rosario
  - AR302, Santa Fe
  - AR306, Santiago del Estero
- Belgium (5):
  - BE003, Bruges
  - BE002, Brussels
  - BE004, Brussels
  - BE005, Leuven
  - BE001, Roeselare
- Brazil (8):
  - BR307, Curitiba
  - BR309, Curitiba
  - BR303, Porto Alegre
  - BR301, Rio de Janeiro
  - BR306, Rio de Janeiro
  - BR302, São Paulo
  - BR304, São Paulo
  - BR308, São Paulo
- Bulgaria (6):
  - BG005, Plovdiv
  - BG001, Sofia
  - BG002, Sofia
  - BG003, Sofia
  - BG004, Sofia
  - BG006, Sofia
- Canada (12):
  - CA002, Gatineau
  - CA309, Gatineau
  - CA301, Halifax
  - CA302, Kelowna
  - CA006, London
  - CA306, Montreal
  - CA008, Newmarket
  - CA304, Qubec
  - CA001, Toronto
  - CA305, Toronto
  - CA308, Toronto
  - CA307, Verdun
- Chile (5):
  - CL004, Antofagasta
  - CL002, Santiago
  - CL003, Santiago
  - CL005, Santiago
  - CL001, Valdivia
- Croatia (3):
  - HR304, Zabok
  - HR301, Zagreb
  - HR302, Zagreb
- Czechia (13):
  - CZ006, Brno
  - CZ309, Choceň
  - CZ306, Hradec Králové
  - CZ007, Kutná Hora
  - CZ004, Pardubice
  - CZ001, Prague
  - CZ002, Prague
  - CZ003, Prague
  - CZ301, Prague
  - CZ303, Prague
  - CZ304, Prague
  - CZ310, Praha 10 - Strasnice
  - CZ005, Rychnov nad Kněžnou
- Denmark (2):
  - DK003, Aarhus N
  - DK001, Copenhagen
- Estonia (3):
  - EE301, Tallinn
  - EE303, Tallinn
  - EE302, Tartu
- Finland (3):
  - FI302, Kuopio
  - FI303, Oulu
  - FI301, Turku
- France (17):
  - FR006, Besançon
  - FR301, Bordeaux
  - FR308, Bron
  - FR309, Élancourt
  - FR008, Limoges
  - FR302, Marseille
  - FR003, Nantes
  - FR312, Nantes
  - FR303, Nice
  - FR001, Paris
  - FR005, Paris
  - FR311, Paris
  - FR306, Reims
  - FR305, Rouen
  - FR004, Saint-Priest-en-Jarez
  - FR313, Saint-Priest-en-Jarez
  - FR002, Toulouse
- Germany (7):
  - DE002, Berlin
  - DE006, Ellwangen
  - DE005, Hanover
  - DE007, Heidelberg
  - DE009, München
  - DE008, Ulm
  - DE004, Unterhaching
- Hungary (4):
  - HU304, Budapest
  - HU305, Budapest
  - HU301, Esztergom
  - HU302, Szeged
- Israel (3):
  - IL302, Haifa
  - IL303, Holon
  - IL304, Ramat Gan
- Italy (18):
  - IT004, Ancona
  - IT006, Brescia
  - IT306, Brescia
  - IT309, Brescia
  - IT313, Cefalù
  - IT002, Florence
  - IT311, Genova
  - IT003, Lamezia Terme
  - IT001, Milan
  - IT312, Monza
  - IT005, Palermo
  - IT007, Palermo
  - IT307, Perugia
  - IT301, Pisa
  - IT305, Roma
  - IT308, Roma
  - IT304, Torino
  - IT310, Torrette
- Lithuania (4):
  - LT302, Kaunas
  - LT303, Kaunas
  - LT301, Vilnius
  - LT304, Vilnius
- Poland (17):
  - PL301, Bialystok
  - PL304, Bydgoszcz
  - PL308, Gdynia
  - PL004, Gliwice
  - PL007, Katowice
  - PL309, Krakow
  - PL302, Lodz
  - PL310, Lubin
  - PL306, Lublin
  - PL307, Oświęcim
  - PL303, Poznan
  - PL005, Późna
  - PL006, Sopot
  - PL002, Szczecin
  - PL311, Szczecin
  - PL003, Warsaw
  - PL008, Wroclaw
- Portugal (2):
  - PT301, Amadora
  - PT302, Coimbra
- Romania (2):
  - RO002, Bucharest
  - RO001, Târgu Mureş
- South Africa (6):
  - ZA003, Bloemfontein
  - ZA006, Cape Town
  - ZA007, Cape Town
  - ZA004, George
  - ZA001, Pretoria
  - ZA002, Rosebank
- South Korea (9):
  - KR303, Busan
  - KR301, Incheon
  - KR308, Seongnam-si
  - KR302, Seoul
  - KR304, Seoul
  - KR305, Seoul
  - KR306, Seoul
  - KR307, Seoul
  - KR309, Seoul
- Spain (6):
  - ES006, Barcelona
  - ES001, Donostia / San Sebastian
  - ES005, Manresa
  - ES004, Salamanca
  - ES002, San Vicent del Raspeig
  - ES003, Santiago de Compostela
- Taiwan (3):
  - TW301, Kaohsiung City
  - TW302, Kaohsiung City
  - TW303, Tainan
- Ukraine (5):
  - UA008, Dnipropetrovsk
  - UA006, Kherson
  - UA005, Kyiv
  - UA007, Kyiv
  - UA001, Lviv
- United Kingdom (11):
  - GB307, Amersham
  - GB301, Glasgow
  - GB303, London
  - GB308, London
  - GB310, London
  - GB306, Plymouth
  - GB311, Plymouth
  - GB309, Prescot
  - GB305, Preston
  - GB304, Southampton
  - GB302, Swindon

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Open-label extension study in patients with mild to moderate AD who completed the 24-week lead-in study 14861A (NCT01955161) or 14862A (NCT02006641)
Groups:
- Idalopirdine 60 mg: Idalopirdine 60 mg adjunct to 10 mg donepezil. The dose of idalopirdine could be decreased from 60 mg to 30 mg if 60 mg was not well tolerated. The dose of donepezil was to be maintained throughout the study.
Period: OLEX
Arm/Group | Idalopirdine 60 mg | Idalopirdine 60 mg + Memantine
Started | 1463 | 0
Completed | 1235 | 0
Not Completed | 228 | 0
Not completed — Withdrawal before treatment | 1 | 0
Not completed — Death | 11 | 0
Not completed — Adverse Event | 66 | 0
Not completed — Withdrawal by Subject | 60 | 0
Not completed — Lost to Follow-up | 6 | 0
Not completed — Protocol Violation | 6 | 0
Not completed — Lack of Efficacy | 3 | 0
Not completed — Results of the lead-in studies | 58 | 0
Not completed — Other: Disallowed medication | 8 | 0
Not completed — Other: Insufficient compliance | 2 | 0
Not completed — Other: Caregiver unavailable | 3 | 0
Not completed — Other: Coordinator decision | 1 | 0
Not completed — Other: Worsening of condition | 1 | 0
Not completed — Other: Moved to nursing home | 1 | 0
Not completed — Other: Withdrawal of caregiver consent | 1 | 0
Period: OLEX-MEM
Arm/Group | Idalopirdine 60 mg | Idalopirdine 60 mg + Memantine
Started | 0 | 101
Completed | 0 | 82
Not Completed | 0 | 19
Not completed — Adverse Event | 0 | 6
Not completed — Withdrawal by Subject | 0 | 7
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other: Moved to nursing home | 0 | 3

BASELINE CHARACTERISTICS:
Population: A total of 1463 patients were enrolled into the study but 1 patient was not treated (did not receive IMP). The baseline analysis population only consist of patients who have been treated. The baseline measures are those collected at entry into the lead-in studies (Baseline I).
Arm/Group | Idalopirdine 60 mg
Number analyzed (Participants) | 1462
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 922
  Male | 540
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 209
  Unknown or Not Reported | 1224
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Information has not been collected
  Asian | 63
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 17
  White | 1318
  More than one race | NA — Information has not been collected
  Unknown or Not Reported | 62
Region of Enrollment [Number; unit: participants]
  Czechia | 135
  United States | 236
  Portugal | 12
  South Korea | 40
  Brazil | 30
  Poland | 139
  Bulgaria | 52
  Chile | 79
  France | 71
  Lithuania | 34
  Croatia | 11
  Argentina | 119
  Romania | 6
  Hungary | 10
  Ukraine | 47
  United Kingdom | 66
  Spain | 50
  Canada | 51
  Belgium | 13
  Finland | 13
  Taiwan | 15
  Denmark | 11
  Italy | 82
  South Africa | 39
  Israel | 5
  Germany | 52
  Estonia | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) in the OLEX
Description: A TEAE is an adverse event that starts or increases in intensity after the date of Baseline II.
Time Frame: Baseline II (start of OLEX, week 0) to end of OLEX (week 28)
Population: All patients who took at least one dose of IMP in the OLEX.
Measure: Number; unit: TEAEs
Arm/Group | Idalopirdine 60 mg
Number analyzed (Participants) | 1462
TEAEs | 2130

2. Primary Outcome: Number of TEAEs in the OLEX-MEM
Description: A TEAE is an adverse event that starts or increases in intensity after the date of Baseline III (start of OLEX-MEM).
Time Frame: From Baseline III (start of OLEX-MEM, Week 28) to end of OLEX-MEM (Week 52)
Population: All patients who took at least one dose of IMP or memantine in the OLEX-MEM.
Measure: Number; unit: TEAEs
Arm/Group | Idalopirdine 60 mg + Memantine
Number analyzed (Participants) | 101
TEAEs | 93

3. Secondary Outcome: Change in Cognition
Description: Change from Baseline II to Week 28 in Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) total score. The ADAS-cog is a 11-item neuropsychological test that assess the severity of cognitive impairment. The items determine the patient's orientation, memory, language, and praxis. Total score of the 11 items range from 0 to 70 (lower score indicates lower cognitive impairment).
Time Frame: Baseline II (start of OLEX, Week 0) to Week 28
Population: All patients in who took at least one dose of IMP in the OLEX.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14681A: Idalopirdine 60 mg adjunct to 10 mg donepezil. The dose of idalopirdine could be decreased from 60 mg to 30 mg if 60 mg was not well tolerated. The dose of donepezil was to be maintained throughout the study.
  Patients from lead-in Study 14681A
- Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14862A: Idalopirdine 60 mg adjunct to 10 mg donepezil. The dose of idalopirdine could be decreased from 60 mg to 30 mg if 60 mg was not well tolerated. The dose of donepezil was to be maintained throughout the study.
  Patients from lead-in Study 14682A
Arm/Group | Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14681A | Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14862A
Number analyzed (Participants) | 693 | 602
units on a scale | 3.01 (0.22) | 2.67 (0.23)

4. Secondary Outcome: Clinical Global Impression Score
Description: Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) score at Week 28. The ADCS-CGIC is a semi-structured interview to assess clinically relevant changes in patients with AD. The items determine cognition, behavior, social and daily functioning. Severity at baseline is rated on a 7-point scale from 1 (normal, not ill at all) to 7 (among the most extremely ill patients). The clinically relevant change from baseline is rated on a 7-point scale from 1 (marked improvement) to 7 (marked worsening).
Time Frame: Week 28
Population: All patients in who took at least one dose of IMP in the OLEX.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14681A | Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14862A
Number analyzed (Participants) | 693 | 594
units on a scale | 4.58 (0.005) | 4.61 (0.05)

5. Secondary Outcome: Change in Daily Functioning
Description: Change from Baseline II to Week 28 in Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL23) total score. The ADCS-ADL23 is a 23-item clinician-rated inventory to assess activities of daily living (conducted with a caregiver or informant). Each item comprises a series of hierarchical sub-questions, ranging from the highest level of independent performance to a complete loss for each activity. Total score of the 23 items ranges from 0 to 78 (higher score indicates lower disability).
Time Frame: Baseline II (start of OLEX, Week 0) to Week 28
Population: All patients in who took at least one dose of IMP in the OLEX.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14681A | Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14862A
Number analyzed (Participants) | 696 | 601
units on a scale | -3.71 (0.28) | -3.88 (0.32)

6. Secondary Outcome: Change in Behavioural Disturbance
Description: Change from Baseline II to Week 28 in Neuropsychiatric Inventory (NPI) total score. The NPI is a 12-item structured interview with a caregiver to assess behavioural disturbances. The NPI comprises 10 behavioural and 2 neurovegetative items. Each item consists of a screening question and several sub-questions that are rated no (not present) or yes (present). Each item is rated for frequency (a 4-point scale from 1 [occasionally] to 4 [very frequent]) and severity (a 3-point scale from 1 [mild] to 3 [marked]). The total NPI score is the frequency ratings multiplied by the severity ratings and ranges from 0 to 144 (higher score indicates worse outcome).
Time Frame: Baseline II (start of OLEX, Week 0) to Week 28
Population: All patients in who took at least one dose of IMP in the OLEX.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14681A | Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14862A
Number analyzed (Participants) | 697 | 602
units on a scale | 1.80 (0.35) | 1.36 (0.34)

7. Secondary Outcome: Change in Cognitive Aspects of Mental Function
Description: Change from Baseline II to Week 28 in Mini Mental State Examination (MMSE). The MMSE is an 11-item test to assess the cognitive aspects of mental function. The subtests assess orientation, memory, attention, language, and visual construction. The scores for each item is dichotomous (1 = response is correct, 0 = response is incorrect). Total score of the 11 items ranges from 0 to 30 (higher score indicates lower deficit).
Time Frame: Baseline II (start of OLEX, Week 0) to Week 28
Population: All patients in who took at least one dose of IMP in the OLEX.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14681A | Idalopirdine 60 mg (OLEX); Patients From lead-in Study 14862A
Number analyzed (Participants) | 730 | 646
units on a scale | -1.28 (0.10) | -1.02 (0.11)

8. Secondary Outcome: Change in Cognitive Aspects of Mental Function
Description: Change from Baseline III to Week 52 in Mini Mental State Examination (MMSE). The MMSE is an 11-item test to assess the cognitive aspects of mental function. The subtests assess orientation, memory, attention, language, and visual construction. The scores for each item is dichotomous (1 = response is correct, 0 = response is incorrect). Total score of the 11 items ranges from 0 to 30 (higher score indicates lower deficit).
Time Frame: Baseline III (start of OLEX-MEM, Week 28) to Week 52
Population: All patients who took at least one dose of IMP or memantine in the OLEX-MEM.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Idalopirdine 60 mg + Memantine (OLEX-MEM): Idalopirdine 60 mg as adjunct to 10 mg donepezil and memantine (patient's individualised maintenance dose, either immediate-release (IR) 20 mg/day (recommended target dose) or extended release (XR) 28 mg/day (recommended target dose). Memantine was administered to approximately 100 patients included in the OLEX-MEM. The dose of idalopirdine could be decreased from 60 mg to 30 mg if 60 mg was not well tolerated. The dose of donepezil was to be maintained throughout the study. The dose of memantine could be changed at any time throughout the study.
Arm/Group | Idalopirdine 60 mg + Memantine (OLEX-MEM)
Number analyzed (Participants) | 93
units on a scale | -0.55 (0.26)

ADVERSE EVENTS:
Time Frame: From Baseline II (week 0) to week 28 (week 32, including safety follow-up, for patients who did not continue in OLEX-MEM) for OLEX. From Baseline III (week 28) to week 56 (including safety follow-up) for OLEX-MEM.
Description: Treatment-Emergent Adverse Events are reported in this section
Arm/Group | Idalopirdine 60 mg | Idalopirdine 60 mg + Memantine
All-Cause Mortality (participants affected / at risk) | 11/1462 | 0/101
Serious Adverse Events (participants affected / at risk) | 91/1462 | 2/101
Other Adverse Events (participants affected / at risk) | 182/1462 | 7/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Idalopirdine 60 mg (N=1462) | Idalopirdine 60 mg + Memantine (N=101)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Iris adhesions (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Retinopathy proliferative (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Exercise tolerance decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 1 | 0
Hepatitis e (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 2 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Pneumonia bacterial (Infections and infestations) | 4 | 0
Septic shock (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 2 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of cervix uteri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/922 | 0/69
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Dementia alzheimer's type (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0
Loss of consciousness (Nervous system disorders) | 2 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Device malfunction (Product Issues) | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Aggression (Psychiatric disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 2 | 0
Delusion (Psychiatric disorders) | 1 | 0
Depressive symptom (Psychiatric disorders) | 1 | 0
Grief reaction (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/540 | 0/32
Breast mass (Reproductive system and breast disorders) | 1 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Social stay hospitalisation (Social circumstances) | 0 | 1
Cataract operation (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idalopirdine 60 mg (N=1462) | Idalopirdine 60 mg + Memantine (N=101)
Accidental overdose (Injury, poisoning and procedural complications) | 105 | 6
Fall (Injury, poisoning and procedural complications) | 80 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-06-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT02079246/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT02079246/SAP_001.pdf